CLINICAL TRIAL: NCT02601092
Title: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic Mini Gastric Bypass: A Randomized Controlled Trial
Brief Title: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic Mini Gastric Bypass
Acronym: MGB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Marko Kraljevic, MD, MD, Spital Limmattal Schlieren
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLS-002
Record Dates: First submitted 2015-09-28; First posted 2015-11-10 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Bypass Complications
Keywords: Mini Gastric Bypass; Roux-en-Y Gastric Bypass; RCT
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini Gastric Bypass (Experimental): The mini gastric bypass procedure was first developed by Dr Robert Rutledge from the USA in 1997, as a modification of the standard Billroth II procedure. A mini gastric bypass creates a long narrow tube of the stomach along its right border (the lesser curvature). A loop of the small gut is brought up and hooked to this tube at about 180 cm from the start of the intestine.
  No drugs or devices will be used.
  Interventions: Procedure: Mini Gastric Bypass
- Roux-en-Y Gastric Bypass (Active Comparator): This variant is the most commonly employed gastric bypass technique, and is by far the most commonly performed bariatric procedure in the United States. The small intestine is divided approximately 45 cm (18 in) below the lower stomach outlet and is re-arranged into a Y-configuration, enabling outflow of food from the small upper stomach pouch via a "Roux limb". In the proximal version, the Y-intersection is formed near the upper (proximal) end of the small intestine. The Roux limb is constructed using 80-150 cm (31-59 in) of the small intestine, preserving the rest (and the majority) of it for absorbing nutrients.
  No drugs or devices will be used.
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Mini Gastric Bypass — The mini gastric bypass procedure was first developed by Dr Robert Rutledge from the USA in 1997, as a modification of the standard Billroth II procedure. A mini gastric bypass creates a long narrow tube of the stomach along its right border (the lesser curvature). A loop of the small gut is brought up and hooked to this tube at about 180 cm from the start of the intestine.
  No drugs or devices will be used.
  Arms: Mini Gastric Bypass
Procedure: Roux-en-Y Gastric Bypass — This variant is the most commonly employed gastric bypass technique, and is by far the most commonly performed bariatric procedure in the United States. The small intestine is divided approximately 45 cm (18 in) below the lower stomach outlet and is re-arranged into a Y-configuration, enabling outflow of food from the small upper stomach pouch via a "Roux limb". In the proximal version, the Y-intersection is formed near the upper (proximal) end of the small intestine. The Roux limb is constructed using 80-150 cm (31-59 in) of the small intestine, preserving the rest (and the majority) of it for absorbing nutrients.
  No drugs or devices will be used.
  Arms: Roux-en-Y Gastric Bypass

SUMMARY:
Several retrospective studies have shown same efficiency in regard to weight loss, with a lower rate of complications for the laparoscopic mini gastric bypass (LMGB) compared to Roux-en-Y gastric bypass (LRYGB). The aim of this double-blinded randomized controlled trial is to compare the two procedures in respect of excess weight loss, complications, operation time, length of stay and the metabolic impact on the hormonal brain-gut-axis.

DETAILED DESCRIPTION:
Bariatric surgery, the only effective treatment for morbid obesity, has shown effective long term weight loss and good control of obesity related comorbidities in randomized controlled trials.

Obesity related diseases, such as hypertension, type 2 diabetes, dyslipidemia, osteoarthritis and various tumours, have a significant socio-economic impact, since the cost of the obesity epidemic is 5.7 billion Swiss francs yearly.

According to the current Swiss National Guidelines defined by the Swiss Group for Morbid Obesity surgical therapy is indicated in cases of BMI 35 kg/m2 or higher, showing better weight reduction and control of comorbidties than conservative therapy alone. Obesity reduces quality of life and life expectancy dramatically. Furthermore it has a significant impact on our economy. Bariatric surgery is likely to improve all of these negative impacts on society.

The most commonly performed procedures at present are laparoscopic adjustable gastric banding, laparoscopic Roux-en-Y gastric bypass (LRYGB) and laparoscopic sleeve gastrectomy (LSG).

LRYGB is considered the golden standard in bariatric surgery, although little evidence is available to justify this standpoint. In fact, the choice of the surgical procedure depends more on patient factors such as present comorbidities and operative risk. Therefore, surgeons consult after a work up within a multidisciplinary team of caretakers such as nutritionists, endocrinologists and psychiatrists and chose a patient tailored approach. Recently, the laparoscopic mini gastric bypass (LMGB) has gained worldwide popularity in addition to the standard available procedures for the treatment of morbid obesity. Therefore, it has been added by the Swiss Group for Morbid Obesity as a surgical option, which has to be evaluated in clinical trials.

Robert Rutledge, the pioneer of the LMGB, published in 2001 results of 1274 patients, who received surgical treatment with LMGB. After two years the patients showed an excess weight loss (EWL) of 77%. The rate of anastomotic leakage in the gastroenterostomy amounted 1.6%. The rate of mortality was 0.08%. Subsequently, Rutledge published in 2005 the results of 2410 patients with a follow up of 38.7 months. These cohort reached/achieved an EWL of 80% after a year and even after 5 years 5% of all these patients showed a weight rebound of maximum 10 kg. In fact, those results seemed superior to outcomes of the other standard bariatric procedures.

The rate of anastomotic leakage was 1.08%, mortality 0.08%. Long-term complications were ulcer disease (4%) and iron deficiency (5%). Both complications are also known in LRYGB with similar rates.

The first and only randomized controlled trial comparing the LRYGB to LMGB was carried out by Lee in 2005. With a group of 40 patients the effectiveness of LMGB was compared to the LRYGB. The authors found an EWL of 64.9% after one and 64.4% after two years, respectively, in patients having a LMGB accompanied by less complications and a shorter hospitalization time than in LRYGB. Patients with LRYGB had an EWL of 58.7% and 60%, respectively.

These results showed similar benefits of the LMGB compared to LRYGB. This is in accordance with the already mentioned observational studies.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* age > 18

Exclusion Criteria:

* malignancy
* lack of compliance
* BMI > 50

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Excess Weight Loss | 1 year postoperative

SECONDARY OUTCOMES:
Early surgical complications | ≤ 30 days
Early non-surgical complications | ≤ 30 days
Operation time | intraoperative
  Operation time measured in minutes for the primary procedure (e.g. LRYGB or LMGB)
Length of stay | up to 24 weeks
  Length of stay after the primary operation (e.g. LRYGB or LMGB)
Subjective perception of the appetite and saturation | 6 weeks, 1 and 3 years
  measured by questionnaires
Hormonal assay (Ghrelin) | preoperative, 6 weeks, 1 and 3 years
  measured in pg/ml
Hormonal assay (GLP-1) | preoperative, 6 weeks, 1 and 3 years
  measured in pg/ml
Hormonal assay (PYY) | preoperative, 6 weeks, 1 and 3 years
  measured in pg/ml
Glucose homeostasis | preoperative, 6 weeks, 1 and 3 years
Lipid profile | preoperative, 6 weeks, 1 and 3 years
  LDL (mg/dl), HDL (mg/dl), triglycerides (mg/dl), total cholesterol (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, MD, Principal Investigator — Spital Limmattal Schlieren
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Result] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Result] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982
- [Result] Rutledge R. The mini-gastric bypass: experience with the first 1,274 cases. Obes Surg. 2001 Jun;11(3):276-80. doi: 10.1381/096089201321336584. PMID 11433900
- [Result] Lee WJ, Yu PJ, Wang W, Chen TC, Wei PL, Huang MT. Laparoscopic Roux-en-Y versus mini-gastric bypass for the treatment of morbid obesity: a prospective randomized controlled clinical trial. Ann Surg. 2005 Jul;242(1):20-8. doi: 10.1097/01.sla.0000167762.46568.98. PMID 15973097
- [Result] Rutledge R, Walsh TR. Continued excellent results with the mini-gastric bypass: six-year study in 2,410 patients. Obes Surg. 2005 Oct;15(9):1304-8. doi: 10.1381/096089205774512663. PMID 16259892
- [Result] Lee WJ, Ser KH, Lee YC, Tsou JJ, Chen SC, Chen JC. Laparoscopic Roux-en-Y vs. mini-gastric bypass for the treatment of morbid obesity: a 10-year experience. Obes Surg. 2012 Dec;22(12):1827-34. doi: 10.1007/s11695-012-0726-9. PMID 23011462
- [Result] Wittgrove AC, Clark GW. Laparoscopic gastric bypass, Roux-en-Y- 500 patients: technique and results, with 3-60 month follow-up. Obes Surg. 2000 Jun;10(3):233-9. doi: 10.1381/096089200321643511. PMID 10929154
- [Result] Rutledge R. Similarity of Magenstrasse-and-Mill and Mini-Gastric bypass. Obes Surg. 2003 Apr;13(2):318. doi: 10.1381/096089203764467315. No abstract available. PMID 12740148
- [Result] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- [Derived] Delko T, Kraljevic M, Lazaridis II, Kostler T, Jomard A, Taheri A, Lutz TA, Osto E, Zingg U. Laparoscopic Roux-Y-gastric bypass versus laparoscopic one-anastomosis gastric bypass for obesity: clinical & metabolic results of a prospective randomized controlled trial. Surg Endosc. 2024 Jul;38(7):3875-3886. doi: 10.1007/s00464-024-10907-7. Epub 2024 Jun 3. PMID 38831218
- [Derived] Kraljevic M, Delko T, Kostler T, Osto E, Lutz T, Thommen S, Droeser RA, Rothwell L, Oertli D, Zingg U. Laparoscopic Roux-en-Y gastric bypass versus laparoscopic mini gastric bypass in the treatment of obesity: study protocol for a randomized controlled trial. Trials. 2017 May 22;18(1):226. doi: 10.1186/s13063-017-1957-9. PMID 28532499